CLINICAL TRIAL: NCT06125106
Title: Prospective, Single-arm, Multicenter Clinical Study on Haploidentical Hematopoietic Stem Cell Transplantation in Patients With MRD Positive CD19+ALL Treated With Conditioning Regimens Containing Blinatumomab
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, He Huang, The President of The First Affiliated Hospital, College of Medicine, Zhejiang University, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT20230044C-R1
Record Dates: First submitted 2023-11-05; First posted 2023-11-09 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-10

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: Minimal Residual Disease; Allogeneic hematopoietic stem cell transplantation; Blinatumomab
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Neoplasm, Residual | interventions — blinatumomab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Blinatumomab Group (Experimental): Haploidentical hematopoietic stem cell transplantation was performed using a Conditioning regimen containing Blinatumomab. 28ug of Blinatumomab was administered intravenously once a day for a total of 7 days, followed by a routine conditioning regimen and haploid hematopoietic stem cell transplantation.
  Interventions: Drug: Blinatumomab

INTERVENTIONS:
Drug: Blinatumomab — Haploidentical hematopoietic stem cell transplantation was performed using a Conditioning regimen containing Blinatumomab. 28ug of Blinatumomab was administered intravenously once a day for a total of 7 days, followed by a routine conditioning regimen and haploid hematopoietic stem cell transplantation.
  Other Names: HSCT

SUMMARY:
A study on the effectiveness and safety of haploidentical hematopoietic stem cell transplantation in patients with MRD positive CD19+ ALL treated with conditioning regimens containing Blinatumomab

DETAILED DESCRIPTION:
This is a prospective multicenter clinical study. This study is applicable to CD19+ ALL patients undergoing allogeneic hematopoietic stem cell transplantation. The purpose is to evaluate the effectiveness and safety of haploidentical hematopoietic stem cell transplantation in patients with MRD positive CD19+ ALL treated with conditioning regimens containing Blinatumomab.31 patients will be included in the study. Clinical endpoints include progress-free survival, Overall survival, cumulative incidence of relapse, non-relapse mortality, minimal residual disease, and graft versus host disease.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed as acute B-ALL with CD19+ according to the 2022 WHO classification criteria. After induction and intensified chemotherapy, complete hematological remission was achieved, but MRD was positive by flow cytometry;
2. Age range from 18 to 70 years old, regardless of gender;
3. The Eastern Oncology Collaborative Group (ECOG) physical fitness score is 0-2 points;
4. Female patients of childbearing age who had a negative pregnancy test before the trial and agreed to take effective contraceptive measures during the trial until their last visit;
5. Organ function is normal, and the following laboratory indicators are met within one week of enrollment: creatinine clearance rate ≥ 60 mL/min (according to the Cockcroft Fault formula); AST and ALT ≤ 3 × Upper limit of normal value range (ULN), total bilirubin ≤ 2 × ULN; Echocardiography (ECHO) shows left ventricular ejection fraction (LVEF) ≥ 50%;
6. Life expectancy greater than 8 weeks;
7. Voluntarily sign an informed consent form to understand and comply with the requirements of the study.

Exclusion Criteria:

1. Failure to achieve complete hematological remission, including residual extramedullary infiltration;
2. Previously received hematopoietic stem cell transplantation;
3. Received systemic chemotherapy within 2 weeks;
4. Previously received treatment with Blinatumomab;
5. Have a history of central nervous system leukemia or present with central nervous system leukemia;
6. Active autoimmune diseases, such as SLE, rheumatoid arthritis, etc;
7. Currently suffering from clinically significant active cardiovascular diseases, such as uncontrolled arrhythmia, uncontrolled hypertension, congestive heart failure, any grade 3 or 4 heart disease determined according to the New York Heart Association (NYHA) functional classification (see Appendix 1), or having a history of myocardial infarction within 6 months prior to screening;
8. Chronic obstructive pulmonary disease with whole lung dysfunction;
9. Other serious diseases that may restrict patients from participating in this test (such as advanced infection, uncontrollable diabetes);
10. Concomitant arteriovenous thrombosis or hypercoagulable state;
11. Known human immunodeficiency virus (HIV) infection, or chronic infection of hepatitis B virus (HBsAg positive) or hepatitis C virus (anti-HCV positive) beyond drug control;
12. Pregnant or lactating women;
13. Severe allergies to other monoclonal antibodies in the past;
14. Those who are unable to understand, comply with the research protocol or sign an informed consent form.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2023-11-16 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Progress-Free Survival | At Year 1
  Progression-free survival (PFS) is defined as the time from transplantation to disease progression or death from any cause.

SECONDARY OUTCOMES:
Overall Survival | At Year 1
  Overall survival (OS) is defined as the time from transplantation to death
Cumulative Incidence of Relapse | At Year 1
  The time from the date of transplantation to disease recurrence:
  Disease recurrence, defined as one of the following:
  Leukemia blasts reappeared in peripheral blood, or blasts ≥ 5%, naive monocytes ≥ 5% in bone marrow, or extramedullary lesions.
Non-relapse Mortality | At Year 1
  NRM was defined as death after transplant that was not preceded by recurrent or progressive malignancy.
Minimal Residual Disease | At Year 1
  Minimal residual disease is a small number of cancer cells left in the body after treatment.
acute graft versus host disease | At Day 100
  assessment of acute GVHD
chornic graft versus host disease | At Year 1
  assessment of chronic GVHD

CONTACTS AND LOCATIONS:
Locations (1):
- The first affiliated hospital of medical college of zhejiang university, Hangzhou, Zhejiang, China